CLINICAL TRIAL: NCT02138422
Title: A Double Blind, Placebo Controlled Pivotal Phase III Study Evaluating Xilonix™ in Symptomatic Colorectal Cancer Patients Refractory to Standard Therapy
Brief Title: A Phase 3 Study to Evaluate Xilonix as an Anticancer Therapy in Patients With Symptomatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-PT026
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Symptomatic Colorectal Cancer; Advanced Colorectal Cancer; Colorectal Cancer With Cachexia
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — bermekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered intravenously every 2 weeks
  Interventions: Biological: Placebo
- Xilonix (Active Comparator): Xilonix administered intravenously every 2 weeks
  Interventions: Biological: Xilonix

INTERVENTIONS:
Biological: Xilonix
  Arms: Xilonix
Biological: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study will be to assess how effective Xilonix is in the treatment of patients with symptomatic colorectal cancer. By blocking a substance that helps tumours grow and spread, Xilonix therapy may not only slow tumour growth, but also may improve symptoms of muscle loss, fatigue, appetite loss, and pain in patients with colorectal cancer. The effectiveness of the therapy will be measured by assessing the change in these symptoms for patients treated with Xilonix versus those treated with placebo. Reversal of muscle loss will be assessed with a type of X-ray called a DEXA scanner. Improvement in pain, appetite loss, and fatigue will be measured with a questionnaire that is completed by patients enrolled on the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with pathologically confirmed colorectal carcinoma that is metastatic or unresectable and which is refractory to standard therapy. To be considered refractory, a subject must have failed both an oxaliplatin (oxaliplatin may have been in the adjuvant setting) and an irinotecan based regimen.
2. Symptomatic Disease: One symptom from each domain (metabolic and functional) must be present.

   * Evidence of metabolic dysfunction, defined as the presence of one or more of the following:
   * Any degree (up to 20%) of unintentional total body weight loss in the previous 6 months
   * Serum Interleukin 6 levels ≥10 pg/ml
   * Evidence of reduced function or presence of cancer related symptoms as determined by EORTC QLQ-C30.
   * Appetite reduction, with a score of >10
   * Presence of fatigue, with a score of >10
   * Presence of Pain, with a score of >10
   * Decreased Role, Emotional and Social function, with a score of < 90.
3. Eastern Cooperative Oncology Group (ECOG) performance status 1 or 2.

Exclusion Criteria:

1. Mechanical obstruction that would prevent adequate oral nutritional intake.
2. >20% total body weight loss in the previous 6 months.
3. Serious uncontrolled medical disorder, or active infection, that would impair the ability of the patient to receive protocol therapy.
4. Uncontrolled or significant cardiovascular disease, including:

   * A myocardial infarction within the past 6 months.
   * Uncontrolled angina within the past 3 months.
   * Congestive heart failure within the past 3 months, if defined as NYHC-II.
   * Diagnosed or suspected congenital long QT syndrome.
   * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, Wolff-Parkinson-White (WPW) syndrome, or torsade de pointes).
   * Any history of second or third degree heart block (may be eligible if currently have a pacemaker).
   * Heart rate < 50 beats per minute on pre-entry electrocardiogram.
   * Uncontrolled hypertension (blood pressure >150 mm Hg systolic and >95 mm Hg diastolic).
5. Dementia or altered mental status that would prohibit the understanding or rendering of informed consent.
6. Subjects who have not recovered from the adverse effects of prior therapy at the time of enrollment to ≤ grade 1; excluding alopecia and grade 2 neuropathy.
7. Subjects who have received extensive prior radiation therapy to the bone marrow. Extensive radiation therapy is defined as treatment of more than one axial bony metastasis. However for subjects with rectal cancer pelvic irradiation, in addition to treatment of one axial bony metastasis, is acceptable.
8. Immunocompromised subjects, including subjects known to be infected with human immunodeficiency virus (HIV).
9. Known hepatitis B surface antigen and/or hepatitis C antibody or known history of infection.
10. History of tuberculosis (latent or active) or positive Interferon-gamma release assay (IGRA).
11. Receipt of a live (attenuated) vaccine within 1 month prior to Randomization
12. Subjects with history of hypersensitivity to compounds of similar chemical or biologic composition to Xilonix™ or any component of its formulations.
13. Women who are pregnant or breastfeeding.
14. WOCBP or men whose sexual partners are WOCBP who are unwilling or unable to use an acceptable method of contraception for at least 1 month prior to randomization, for the duration of the study, and for at least 3 months after the last dose of study medication.
15. History of progressive multifocal leukoencephalopathy or other demyelinating disease.
16. Subjects on immunosuppressive therapy, including transplant patients.
17. Subjects with known brain metastases. Subjects with symptoms of brain metastases during screening should undergo CT imaging prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2014-07-31 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Response Rate | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- XBiotech Investigative Site, Warsaw, Poland

REFERENCES:
- [Background] Hong DS, Hui D, Bruera E, Janku F, Naing A, Falchook GS, Piha-Paul S, Wheler JJ, Fu S, Tsimberidou AM, Stecher M, Mohanty P, Simard J, Kurzrock R. MABp1, a first-in-class true human antibody targeting interleukin-1alpha in refractory cancers: an open-label, phase 1 dose-escalation and expansion study. Lancet Oncol. 2014 May;15(6):656-66. doi: 10.1016/S1470-2045(14)70155-X. Epub 2014 Apr 17. PMID 24746841
- [Result] Hickish T, Andre T, Wyrwicz L, Saunders M, Sarosiek T, Kocsis J, Nemecek R, Rogowski W, Lesniewski-Kmak K, Petruzelka L, Apte RN, Mohanty P, Stecher M, Simard J, de Gramont A. MABp1 as a novel antibody treatment for advanced colorectal cancer: a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2017 Feb;18(2):192-201. doi: 10.1016/S1470-2045(17)30006-2. Epub 2017 Jan 14. PMID 28094194